CLINICAL TRIAL: NCT05285202
Title: Clinic Versus Hotspot Active Case Finding and Linkage to Preventive Therapy (ACF/TPT) Strategy Evaluation for TB: A Cluster-Randomized Crossover Trial
Brief Title: Clinic-based Versus Hotspot-focused Active TB Case Finding
Acronym: CHASE-TB
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH); Walimu (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Screening
Other Study IDs: IRB00300939; 2R01HL138728 (NIH)
Record Dates: First submitted 2022-03-09; First posted 2022-03-17 (Actual); Last update posted 2025-03-04 (Actual); Status verified 2025-02

CONDITIONS: Tuberculosis, Pulmonary; Mycobacterium Tuberculosis Infection
MeSH Terms: conditions — Tuberculosis, Pulmonary; Tuberculosis

STUDY DESIGN:
Intervention Model Description: Twelve clusters or study regions (of which eight will be randomized to receive interventions) will be defined according to the catchment areas of twelve participating Ugandan district hospitals/major health centers. Eight study areas will receive a total of six 4-month intervention periods (alternating between the facility-based and the hotspot focused strategy, for three periods of each type) over a four-year period, with a 4-month wash-out period after each intervention period. Four additional areas will be used as control sites; the only involvement of participants in these sites will be through retrospective collection of de-identified data.
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Hotspot-focused ACF/TPT (Experimental): ACF/TPT intervention will be delivered in a community setting, in geographic areas judged likely to have a high burden of undiagnosed TB
  Interventions: Other: Active TB case finding with linkage to preventive therapy (ACF/TPT)
- Facility-based ACF/TPT (Experimental): ACF/TPT intervention will be delivered on the grounds of a health facility (hospital or large public health center)
  Interventions: Other: Active TB case finding with linkage to preventive therapy (ACF/TPT)
- No intervention (No Intervention)

INTERVENTIONS:
Other: Active TB case finding with linkage to preventive therapy (ACF/TPT) — ACF/TPT in both intervention arms will consist of TB screening by mobile chest X-ray (with artificial intelligence-based reading, followed by confirmatory sputum testing with Xpert MTB/RIF Ultra for participants with abnormal x-rays), and linkage to preventive therapy for those who are TB-negative and eligible for TPT (limited in April 2024 to those with close TB contact or known HIV infection).
  Arms: Facility-based ACF/TPT; Hotspot-focused ACF/TPT

SUMMARY:
This five-year study will evaluate two strategies for conducting tuberculosis (TB) active case finding (ACF) and linkage to TB treatment or TB preventive therapy (TPT) in peri-urban Uganda. The two strategies differ in the location where ACF activities are performed: A "facility-based" ACF/TPT strategy will perform ACF, plus linkage to TPT, in the immediate vicinity of a large public health facility and will primarily recruit individuals who are attending the health facility, irrespective of TB suspicion or symptoms. Alternatively, a "hotspot-based" strategy will use routine notification data and local expertise to identify local TB hotspots - defined as the geographic areas though to have the highest burden of undiagnosed TB per estimated population. The same infrastructure (personnel, equipment, supplies, etc.) for ACF/TPT will then be placed in those zones for a period of four months at a time, and the general population will be recruited for screening and linkage to TPT.

The two interventions will be compared in a Type 1 hybrid effectiveness-implementation trial with a cluster-randomized, multiple-period crossover design. The study will evaluate whether hotspot-focused ACF/TPT results in a greater number of TB patients diagnosed and linked to care, and a greater number of individuals started on preventive therapy, than facility-based ACF/TPT. Secondarily, it will also compare the two interventions in terms of number of people initiated on TPT, and it will compare TB cases detected in regions performing ACF/TPT (either approach) against cases detected in regions that continue to perform the standard of care.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥15 years, OR age 5-14 and a close contact of someone diagnosed with TB,
* Provision of oral informed consent, or, if age <18 years and not legally emancipated, oral informed assent (if ages 8-17) and parental informed consent (ages 5-17) to participate in the study
* Ability to communicate with study staff in English or Luganda, or availability of a capable interpreter who is acceptable to the participant

Exclusion Criteria:

* On treatment for, or diagnosed with but not yet treated for, active TB

Min Age: 5 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 150000 (Estimated)
Dates: Start 2022-06-01 (Actual); Primary Completion 2027-01-31 (Estimated); Study Completion 2027-01-31 (Estimated)

PRIMARY OUTCOMES:
Pulmonary bacteriologically confirmed TB notifications, hotspot vs facility | From the start to two weeks after the end of each four-month intervention period
  Number of study region residents notified as initiating treatment for bacteriologically confirmed new or relapsed pulmonary TB, comparing periods in which regions performed hotspot-focused ACF/TPT to those in which facility-based ACF/TPT was performed.

SECONDARY OUTCOMES:
TPT initiations, hotspot vs facility | From the start to two weeks after the end of each four-month intervention period
  Number of study region residents initiating TPT during intervention periods, comparing periods in which regions performed hotspot-focused ACF/TPT to those in which facility-based ACF/TPT was performed.
Pulmonary bacteriologically confirmed TB notifications, ACF/TPT vs control | 48 months from start of interventions in each "triplet" of clusters
  Number of study region residents notified as initiating treatment for bacteriologically confirmed new or relapsed pulmonary TB, comparing intervention regions to control regions.
Notification trend (intervention vs control) as assessed by Average percent change in number of TB notifications | First 16 months following start of interventions in a cluster "triplet", versus final 16 months of the interventions (including 4 months of washout after the final intervention) in each triplet
  Average percent change in number of TB notifications, from the first 16 months of intervention to the final 16 months of intervention, comparing intervention clusters to control clusters.
Study-initiated TB notifications, hotspot vs facility | From the start to two weeks after the end of each four-month intervention period
  Number of people diagnosed with TB through study participation and initiating treatment for TB, hotspot-focused and facility-based ACF/TPT.
Number screened by study | During four-month intervention periods (6 periods per cluster over 48 months)
  Total number of people screened for TB with each intervention.
Number diagnosed by study | During four-month intervention periods (6 periods per cluster over 48 months)
  Number of study participants found to have Xpert-positive sputum.
Cost effectiveness (hotspot vs facility) as assessed by cost per disability-adjusted life year averted | From the start to two weeks after the end of each four-month intervention period
  Incremental cost per disability-adjusted life year (DALY) averted, comparing the more to the less effective ACF/TPT intervention (if an effectiveness difference is found).
Cost effectiveness (ACF/TPT vs no intervention) as assessed by cost per disability-adjusted life year averted | From the start to two weeks after the end of each four-month intervention period
  Incremental cost per disability-adjusted life year (DALY) averted, comparing ACF/TPT to no ACF/TPT.
Number evaluated for latent tuberculosis infection (LTBI) with tuberculin skin testing (TST) | During four-month intervention periods (6 periods per cluster over 48 months)
  Total number of people completing TST placement and reading by the study
Number referred for TPT | During four-month intervention periods (6 periods per cluster over 48 months)
  Number of participants referred for TB preventive therapy based on TST result or other eligibility criteria
Contacts screened | During four-month intervention periods (6 periods per cluster over 48 months)
  Number of people screened for TB who are identified as contacts of a person diagnosed with TB through the study

CONTACTS AND LOCATIONS:
Overall Officials: Emily Kendall, MD PhD, Principal Investigator — Johns Hopkins University
Locations (1):
- Walimu, Kampala, Uganda

IPD SHARING:
Plan to Share IPD: Yes
Data that underlie results in publications will be deposited into a publicly available data repository at the time of publication.